CLINICAL TRIAL: NCT04011020
Title: Clinical Application of Stem Cell Educator Therapy in Type 1 Diabetes
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Throne Biotechnologies Inc. (Industry)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-TH-002
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Treatment group receive Stem Cell Educator therapy, control group receive conventional insulin therapy.
Who Masked: Care Provider, Investigator
Masking Description: All recruited T1D subjects will receive the treatment with Stem Cell Educator therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment of T1D with Stem Cell Educator therapy (Experimental): Recruited T1D subjects will receive one treatment with SCE therapy.
  Interventions: Combination Product: Stem Cell Educator therapy
- Conventional insulin therapy (Experimental): Control group will receive conventional insulin therapy.
  Interventions: Combination Product: Stem Cell Educator therapy

INTERVENTIONS:
Combination Product: Stem Cell Educator therapy — Patients with T1D will be evaluated by the study principal investigator or co-investigators. Informed consent will be obtained at the initial screening visit. The initial screening visit will occur within 30 days of initiation of SCE therapy. The second screening visit will occur within 7 days of therapy. Subjects who meet all criteria will be scheduled for treatment. All enrolled subjects will receive treatment with the SCE system consisting of a single session of mononuclear cells (MNC) collection by apheresis where 10 L of blood will be processed on day -1. The MNC product will then be exposed over to the SCE and on day 0 the product will be infused intravenously back to the patient.

SUMMARY:
Type 1 diabetes (T1D) is a T cell-mediated autoimmune disease that causes a deficit of pancreatic islet beta cells. Millions of individuals worldwide have T1D, and incidence increases annually. Several recent clinical trials point to the need for an approach that produces comprehensive immune modulation at both the local pancreatic and systemic levels. Stem Cell Educator (SCE) therapy offers comprehensive immune modulation at both the local and systemic levels in T1D by using a patient's own immune cells (including platelets) that are "educated" by cord blood stem cells. Tested clinically in more than 200 patients, SCE therapy has shown lasting reversal in autoimmunity in T1D patients, including improved C-peptide levels, reduced median glycated hemoglobin A1C (HbA1C) values, and decreased median daily usage of insulin. SCE therapy circulates a patient's blood through a blood cell separator, briefly cocultures the patient's immune cells with adherent Cord Blood Stem Cells (CB-SCs) in vitro, and returns the "educated" autologous immune cells to the patient's circulation.

DETAILED DESCRIPTION:
The SCE device is made of a hydrophobic material from FDA-approved (USP Class VI) dishes that tightly binds stem cells CB-SCs without interfering with their immune modulating capability. We originally designed a chamber for co-culture of lymphocytes and CB-SCs that included nine discs of the material with a flow pathway and adherent CB-SCs sandwiched between a top cover plate and a bottom collecting plate. In this trial, we are going to use the 12-layer SCE device.

The SCE therapy carried a lower risk of infection than a typical blood transfusion, and did not introduce stem cells or reagents into the patients. In addition, CB-SCs have very low immunogenicity, and the CB-SCs cultured in the device are a highly restricted population and contain no CD3+ T cells or other lymphocyte subsets, eliminating the need for human leukocyte antigen (HLA) matching prior to treatment. This innovative approach has the potential to provide CB-SC-mediated immune modulation therapy for multiple autoimmune diseases while mitigating the safety and ethical concerns associated with other approaches such as T1D, type 2 diabetes (T2D), and alopecia areata (AA) in clinics. The relative simplicity of the approach may also provide cost and time savings relative to other approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ( 14 years)
2. Must have a diagnosis of type 1 diabetes mellitus based on the 2015 American Diabetes Association criteria for the Clarification and Diagnosis of diabetes.
3. Must have a blood test confirming the presence of at least one autoantibody to pancreatic islet Cells (IAA, IA2, GAD 65, ZnT8).
4. Fasting C-peptide level > 0.3 ng/ml
5. HbA1C < 10% at enrollment
6. Recent diagnosis (within two years of enrollment)
7. Adequate venous access for apheresis
8. Must be equipped with a continuous glucose monitoring system (CGMS)
9. Ability to provide informed consent
10. For female patients only, willingness to use FDA-recommended birth control (http://www.fda.gov/downloads/ForConsumers/ByAudience/ForWomen/FreePublications/UCM356451.pdf) until 6 months post treatment.
11. Must agree to comply with all study requirements and be willing to complete all study visits

Exclusion Criteria:

1. AST or ALT 2 > x upper limit of normal.
2. Abnormal bilirubin (total bilirubin > 1.2 mg/dL, direct bilirubin > 0.4 mg/dL)
3. Creatinine > 2.0 mg/dl.
4. Known coronary artery disease or EKG suggestive of coronary artery disease unless cardiac clearance for apheresis is obtained from a cardiologist.
5. Known active infection such as Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV)
6. Pregnancy assessed by a positive serum pregnancy test or breastfeeding mothers
7. Use of immunosuppressive medication within one month of enrollment including but not limited to prednisone, cyclosporine, tacrolimus, sirolimus, and chemotherapy.
8. Presence of any other autoimmune diseases (lupus, rheumatoid arthritis, scleroderma, etc.)
9. Anticoagulation other than ASA.
10. Hemoglobin < 10 g/dl or platelets < 100 k/ml
11. Is unable or unwilling to provide informed consent
12. Presence of any other physical or psychological medical condition that, in the opinion of the investigator, would preclude participation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Adverse Events in T1D Subjects | 6 month
  The occurrence of treatment-related adverse events will be evaluated post the treatment with SCE therapy.

SECONDARY OUTCOMES:
Preliminary efficacy of SCE therapy to improve beta cell function | 12 months
  Preliminary efficacy as measured by Area under the C-peptide curve (AUC) over the first 2 hours of a 3-hour mixed meal tolerance test (MMTT)
Preliminary efficacy of SCE therapy to improve glucose control | 12 months
  Change in HbA1C levels over time
Preliminary efficacy of SCE therapy to reduce insulin dose | 12 months
  Change in daily insulin requirements
Efficacy of SCE therapy in immune modulation | 12 month
  Measurements of immune markers at baseline, 1, 3, 6, 9, and 12 months. Peripheral blood mononuclear cells (PBMC) will be collected and tested by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: YONG ZHAO, MD,PhD, Study Chair — Throne Biotechnologies Inc.
Locations (2):
- United States (2):
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Throne Biotechnologies, Paramus, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Knight CM, Jiang Z, Delgado E, Van Hoven AM, Ghanny S, Zhou Z, Zhou H, Yu H, Hu W, Li H, Li X, Perez-Basterrechea M, Zhao L, Zhao Y, Giangola J, Weinberg R, Mazzone T. Stem Cell Educator therapy in type 1 diabetes: From the bench to clinical trials. Autoimmun Rev. 2022 May;21(5):103058. doi: 10.1016/j.autrev.2022.103058. Epub 2022 Jan 31. PMID 35108619
- [Result] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Result] Zhao Y. Stem cell educator therapy and induction of immune balance. Curr Diab Rep. 2012 Oct;12(5):517-23. doi: 10.1007/s11892-012-0308-1. PMID 22833322
- [Result] Delgado E, Perez-Basterrechea M, Suarez-Alvarez B, Zhou H, Revuelta EM, Garcia-Gala JM, Perez S, Alvarez-Viejo M, Menendez E, Lopez-Larrea C, Tang R, Zhu Z, Hu W, Moss T, Guindi E, Otero J, Zhao Y. Modulation of Autoimmune T-Cell Memory by Stem Cell Educator Therapy: Phase 1/2 Clinical Trial. EBioMedicine. 2015 Nov 5;2(12):2024-36. doi: 10.1016/j.ebiom.2015.11.003. eCollection 2015 Dec. PMID 26844283
- [Result] Zhao Y, Jiang Z, Delgado E, Li H, Zhou H, Hu W, Perez-Basterrechea M, Janostakova A, Tan Q, Wang J, Mao M, Yin Z, Zhang Y, Li Y, Li Q, Zhou J, Li Y, Martinez Revuelta E, Maria Garcia-Gala J, Wang H, Perez-Lopez S, Alvarez-Viejo M, Menendez E, Moss T, Guindi E, Otero J. Platelet-Derived Mitochondria Display Embryonic Stem Cell Markers and Improve Pancreatic Islet beta-cell Function in Humans. Stem Cells Transl Med. 2017 Aug;6(8):1684-1697. doi: 10.1002/sctm.17-0078. Epub 2017 Jul 7. PMID 28685960
- See also: Throne Biotechnologies Inc — https://thronebio.com/